CLINICAL TRIAL: NCT02678416
Title: A Randomized, Placebo-Controlled, Double-Blind, Two-Part, Cross-over Study in Healthy Adult Male Subjects to Compare the Reduction in Pain Intensity After Single-Dose Administration of Intravenous or Oral Acetaminophen and Intravenous Morphine by Using UVB Burn and Intradermal Capsaicin Experimental Pain Models
Brief Title: Reduction in Pain Intensity Following IV or Oral Pain-relieving Products
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MNK14504055
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-11

CONDITIONS: Pain
Keywords: comparison
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- IV Acetaminophen (Experimental): All participants receive IV acetaminophen as one of 4 interventions in random sequence
  Interventions: Drug: IV Acetaminophen (Treatment A); Drug: Placebo (Treatment C)
- Oral Acetaminophen (Experimental): All participants receive oral acetaminophen as one of 4 interventions in random sequence
  Interventions: Drug: Oral Acetaminophen (Treatment B); Drug: Placebo (Treatment C)
- Placebo (Experimental): All participants receive placebo as one of 4 interventions in random sequence
  Interventions: Drug: Placebo (Treatment C)
- Morphine (Experimental): All participants receive morphine as one of 4 interventions in random sequence
  Interventions: Drug: Placebo (Treatment C); Other: Morphine (Treatment D)

INTERVENTIONS:
Drug: IV Acetaminophen (Treatment A) — Acetaminophen administered by intravenous (IV) infusion
  Other Names: OFIRMEV
  Arms: IV Acetaminophen
Drug: Oral Acetaminophen (Treatment B) — Acetaminophen administered by oral tablets
  Other Names: Acetaminophen tablets
  Arms: Oral Acetaminophen
Drug: Placebo (Treatment C) — Placebo administered by IV infusion or oral tablets
  Other Names: IV Placebo; Placebo tablets
Other: Morphine (Treatment D) — Morphine administered by IV infusion
  Other Names: IV Morphine
  Arms: Morphine

SUMMARY:
The purpose of this study is to evaluate two experimental pain models to see if they would be useful for comparing different products for reduction in pain intensity.

The models evaluated were the ultraviolet-B (UVB) burn and intradermal capsaicin experimental pain models. Medications compared were a single dose each, of intravenous (IV) acetaminophen, oral acetaminophen, placebo, and IV morphine.

ELIGIBILITY:
Inclusion Criteria

1. Must have a health status of "healthy" assessed by the investigator and defined as no clinically significant deviation from normal medical history, physical examination, vital signs, and clinical laboratory determinations.
2. Must be male, Caucasian, between 18 and 55 years of age (inclusive) at the time of the screening.
3. Must have a body mass index (BMI) ≥ 19.0 and ≤ 30.0 kg/m2 with a minimum weight of 110 pounds (50 kg) at screening.

Exclusion Criteria

1. A positive test result for human immunodeficiency virus (HIV), hepatitis B (surface antigen), or hepatitis C virus antibody at Screening.
2. A history of any drug allergy, hypersensitivity, or intolerance to acetaminophen, morphine, or capsaicin or to any of the excipients in the IV or oral formulations used.
3. A positive test result for drugs of abuse, alcohol, or cotinine.
4. Fitzpatrick Skin Type V or VI (based on a Skin Type score of greater than 30.
5. A history of conditions which might be specifically contraindicated or require caution to be used during the administration of any drug in the study.
6. Any other medical, psychiatric and/or social reason for exclusion as determined by the investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-06-13 (Actual); Study Completion 2016-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (1):
- Pharmaceuticals Research Associates, Inc. (PRA), Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 79 participants were enrolled in the study. 12 participants in Part 1 and 66 participants in Part 2 were randomized to sequence, and received at least one dose of the study treatment.
Pre-assignment Details: One participant in Part 2 was randomized but discontinued without receiving treatment due to an adverse event.
Groups:
- Part 1: All participants receive all products in random sequence
Period: Part 1
Arm/Group | Part 1
Started | 12
Safety Population | 12
Modified Intent to Treat (mITT) | 12
Per Protocol Population | 8
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Part 2
Arm/Group | Part 1
Started | 67 (Part 2 enrolled all new participants)
Treated (Safety Population) (One participant was randomized but not treated.) | 66
Modified Intent to Treat Population | 66
Pharmacokinetic Population | 65
Per Protocol Population | 64
Completed | 64
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Population, defined as participants enrolled in the study that received any quantity of study drugs. All new participants were enrolled in Part 2.
Groups:
- Part 1: All participants who received a drug product in Part 1
- Part 2: All participants who received a drug product in Part 2
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 12 | 66 | 78
Age, Continuous [Mean (Full Range); unit: years] | 28.9 [19 to 49] | 26.5 [18 to 52] | 26.9 [18.2 to 51.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 66 | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, White: Not Hispanic or Latino | 12 | 60 | 72
  Race, White: Hispanic or Latino | 0 | 6 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 66 | 78

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline in Pain Intensity at Hour 6 Using the Thermal Suprathreshold Pain in the Ultraviolet-B (UVB) Burn Pain Model
Description: The UVB burn pain model is a validated screening tool for pain killers in clinical drug development. A temperature of 50 degrees centigrade (°C) is used to burn the participant for 5 seconds. Then the participant rates his pain on a scale from 0 (no pain) to 10 (most intense pain). That score is recorded as baseline. Then the participant rates his pain again six hours after taking the assigned medication. The average at baseline is subtracted from the average at hour 6. Because this is a measure of reduction in pain intensity, a higher score is better (it means there is more pain relief).
Time Frame: within 6 hours
Population: Completers, defined as participants who were enrolled in the study, took the entire dose of all study drugs, and provided all pain intensity assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- IV Acetaminophen: All participants received IV acetaminophen
- Oral Acetaminophen: All participants received oral acetaminophen
- Placebo: All participants received placebo
- Morphine: All participants received morphine
Arm/Group | IV Acetaminophen | Oral Acetaminophen | Placebo | Morphine
Number analyzed (Participants) | 11 | 11 | 11 | 11
score on a scale | 0.73 (1.104) | -0.64 (1.804) | -0.36 (1.567) | 0.36 (1.206)

2. Secondary Outcome: Part 2: Observed Thermal Suprathreshold Pain Intensity in the UVB Burn Area
Description: Participants rated their pain intensity on a scale of 0 (no pain) to 10 (most intense pain). The observed mean and standard deviation are disclosed through Hour 6
Time Frame: within 6 hours
Population: Per-Protocol Population, defined as participants who were enrolled in the study, have taken the entire dose of all study drugs, and provided all pain intensity assessments designed for the UVB Burn Pain Model without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Part 2: IV Acetaminophen: All participants received IV acetaminophen
- Part 2: Oral Acetaminophen: All participants received oral acetaminophen
- Part 2: Placebo: All participants received placebo
- Part 2: IV Morphine: All participants received morphine
Arm/Group | Part 2: IV Acetaminophen | Part 2: Oral Acetaminophen | Part 2: Placebo | Part 2: IV Morphine
Number analyzed (Participants) | 64 | 64 | 64 | 64
scores on a scale
  Baseline | 5.4 (1.30) | 5.5 (1.40) | 5.5 (1.32) | 5.6 (1.40)
  0.25 Hours | 5.2 (1.39) | 5.3 (1.48) | 5.5 (1.28) | 4.9 (1.56)
  0.5 Hours | 5.0 (1.34) | 5.1 (1.36) | 5.3 (1.28) | 4.7 (1.50)
  0.75 Hours | 5.0 (1.37) | 5.1 (1.30) | 5.4 (1.26) | 4.7 (1.62)
  1 Hour | 5.0 (1.44) | 4.9 (1.23) | 5.2 (1.34) | 4.6 (1.55)
  2 Hours | 5.3 (1.13) | 5.1 (1.26) | 5.6 (1.28) | 5.1 (1.50)
  3 Hours | 5.4 (1.30) | 5.2 (1.44) | 5.5 (1.23) | 5.0 (1.67)
  4 Hours | 5.5 (1.17) | 5.4 (1.40) | 5.5 (1.30) | 5.2 (1.42)
  6 Hours | 5.6 (1.32) | 5.5 (1.30) | 5.5 (1.34) | 5.4 (1.45)

ADVERSE EVENTS:
Time Frame: From first dose up to Day 46
Description: Safety population included participants enrolled in the study that received any quantity of study medications.
Groups:
- Part 1: IV Acetaminophen; Part 2: IV Acetaminophen: All participants received IV acetaminophen
- Part 1: Oral Acetaminophen; Part 2: Oral Acetaminophen: All participants received oral acetaminophen
- Part 1: Placebo; Part 2: Placebo: All participants received placebo
- Part 1: Morphine; Part 2: Morphine: All participants received morphine
Arm/Group | Part 1: IV Acetaminophen | Part 1: Oral Acetaminophen | Part 1: Placebo | Part 1: Morphine | Part 2: IV Acetaminophen | Part 2: Oral Acetaminophen | Part 2: Placebo | Part 2: Morphine
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/64 | 0/65 | 0/65 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/64 | 0/65 | 0/65 | 0/64
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12 | 4/12 | 8/12 | 10/64 | 12/65 | 14/65 | 38/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: IV Acetaminophen (N=12) | Part 1: Oral Acetaminophen (N=12) | Part 1: Placebo (N=12) | Part 1: Morphine (N=12) | Part 2: IV Acetaminophen (N=64) | Part 2: Oral Acetaminophen (N=65) | Part 2: Placebo (N=65) | Part 2: Morphine (N=66)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 9
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 4 | 1 | 2 | 1 | 20
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 4 | 3 | 4
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 5
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 10
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Axillary Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal Dreams (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Head Discomfort (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Feeling Of Relaxations (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye Movement Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Altered visual depth perception (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators will be part of the primary publication. Each investigator may publish on the data from subjects enrolled at their site after the initial publication has been submitted.